CLINICAL TRIAL: NCT01870843
Title: Improving Quality of Life and Social Functionality With Escitalopram in the Treatment of Major Depressive Disorder With Anxiety Symptom
Brief Title: A Study to Evaluate the Impact of Escitalopram on Quality of Life and Social Functionality in Patients With Major Depressive Disorder With Anxiety Symptom
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Xian-Janssen Pharmaceutical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR100826; ESCITALDEP4005 (Other: Xian-Janssen Pharmaceutical Ltd., China); ESC-C-11-CN-002-V04 (Other: Xian-Janssen Pharmaceutical Ltd., China)
Record Dates: First submitted 2013-06-03; First posted 2013-06-06 (Estimated); Results first posted 2016-07-11 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-05

CONDITIONS: Depressive Disorder, Major
Keywords: Depressive Disorder, Major; Depressive Disorder; Depression; Anxiety; Escitalopram; Quality of life; Social functionality
MeSH Terms: conditions — Depressive Disorder, Major; Depressive Disorder; Depression; Anxiety Disorders | interventions — Escitalopram

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Escitalopram (Experimental): Participants will receive escitalopram 10 mg per day for 1 week and then the dose of escitalopram will be flexibly adjusted up to maximum of 20 mg per day for the next 7 weeks, based on the investigator's clinical judgment.
  Interventions: Drug: Escitalopram

INTERVENTIONS:
Drug: Escitalopram — Escitalopram will be administered as oral tablets 10 mg per day and then the dose of escitalopram will be flexibly adjusted up to maximum of 20 mg per day for the next 7 weeks, based on the investigator's clinical judgment.

SUMMARY:
The purpose of this study is to evaluate the impact of escitalopram on quality of life and social functionality in patients with major depressive disorder with anxiety symptom.

DETAILED DESCRIPTION:
This is an open-label (all people know the identity of the intervention), multi-center, prospective (a study in which the participants are identified and then followed forward in time for the outcome of the study), single-arm (all participants receiving one intervention) study. Approximately 260 participants will be enrolled in this study. This study consists of two phases: screening phase and treatment phase. In the treatment phase, participants will receive escitalopram for 8 weeks: escitalopram 10 mg per day for 1 week and then the dose of escitalopram will be flexibly adjusted up to maximum of 20 mg per day for the next 7 weeks, based on the investigator's clinical judgment. Safety evaluations will include assessment of adverse events, clinical laboratory tests, electrocardiogram, vital signs, and physical examination which will be monitored throughout the study. The total study duration will be approximately 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of major depressive disorder according to the American Psychiatric Association's Diagnostic and Statistical Manual-IV, Text Revision (DSM-IV-TR) diagnostic criteria
* Minimum scores of 9 on Sheehan Disability Scale
* Minimum scores of 14 on Hamilton Anxiety Scale

Exclusion Criteria:

* History of primary or comorbid diagnoses of schizophrenia, schizoaffective disorder, bipolar disorder, or dementia
* Presence of unstable serious illness and/or has a clinically significant renal or hepatic impairment, seizure disorders or any other disease which may be detrimental to the participant or the study
* Participant who have continuously taken psychoactive substances, antidepressants, anxiolytics, Monoamine oxidase inhibitors, psychoactive herbal remedies, lithium, electroconvulsive therapy, carbamazepine in the past 2 weeks before the baseline visit
* Diagnosis of major depressive disorder who currently require treatment systematically within past 2 months from baseline
* Receiving pharmacological treatment, which is disallowed in the current approved Chinese summary of product characteristics for escitalopram

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 261 (Actual)
Dates: Start 2014-03; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Xian-Janssen Pharmaceutical Ltd., China Clinical Trial, Study Director — Xian-Janssen Pharmaceutical Ltd.
Locations (10):
- China (10):
  - Beijing
  - Guangzhou
  - Hangzhou
  - Hohhot
  - Jinan
  - Kunming
  - Nanjing
  - Shijiazhuang
  - Ürümqi
  - Xiamen

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted between 09 April 2014 and 04 May 2015 and recruited participants from 10 study centers in China.
Pre-assignment Details: Of the 261 participants enrolled, 241 participants were included in the Full Analysis Set.
Groups:
- Escitalopram Oxalate: Participants received escitalopram 10 milligram (mg) per day for 1 week and then the dose of escitalopram flexibly adjusted up to maximum of 20 mg per day for the next 7 weeks, based on the investigator's clinical judgment.
Period: Overall Study
Arm/Group | Escitalopram Oxalate
Started | 261
Completed | 208
Not Completed | 53
Not completed — Adverse Event | 10
Not completed — Lost to Follow-up | 24
Not completed — Death | 1
Not completed — Withdrawal by Subject | 18

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS): All randomized participants taking at least one dose of study drug and having at least one visit evaluation in treatment phase were included in the FAS.
Arm/Group | Escitalopram Oxalate
Number analyzed (Participants) | 241
Age, Continuous [Mean (Standard Deviation); unit: Years] — N= 240
  Years | 39.0 (12.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 156
  Male | 85

OUTCOME MEASURES:

1. Primary Outcome: Change in Quality of Life Enjoyment and Satisfaction Questionnaire, Short Form (Q-LES-Q-SF) From Baseline up to Day 56
Description: Q-LES-Q-SF is a 14-item questionnaire in which each question is rated on a 5-point scale with scores ranging from "1 = very poor" to "5 = very good". The total raw score is calculated by summing up the scores for the 14 items. The raw total score ranges from 14 to 70. The raw total score is transformed into a percentage maximum possible score using the following formula: (raw total score minus minimum score) divided by (maximum possible raw score minus minimum score). The minimum raw score on the Q-LES-Q-SF is 14, and the maximum score is 70. Lower score indicate worsening.
Time Frame: Baseline, Day 14, Day 28, Day 42 and Day 56
Population: Full Analysis Set Population included who received at least 1 dose of the study drug, and completed at least 1 assessment visit during the treatment period. Here "n" (Number of Participants Analyzed) signifies number of Participants who were evaluable for this outcome at given time point.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Escitalopram Oxalate
Number analyzed (Participants) | 239
Units on a scale
  Baseline (n=239) | 39.3 (14.43)
  Change at Day 14 (n=219) | 9.6 (15.43)
  Change at Day 28 (n=230) | 15.1 (18.25)
  Change at Day 42 (n=230) | 19.0 (19.56)
  Change at Day 56 (n=230) | 22.5 (20.70)

2. Primary Outcome: Change in Sheehan Disability Scale (SDS) From Baseline up to Day 56
Description: SDS is a composite of 3 self-rated items designed to measure the extent to which 3 major sectors in the participant's life are impaired by panic, anxiety, phobic, or depressive symptoms. The participant rates the extent to which his or her (1) work, (2) social life or leisure activities, and (3) home life or family responsibilities are impaired by his or her symptoms on a 10-point visual analog scale. To get a total score add up the 3 individual scores and the total score ranges from "0 = unimpaired" to "30 = highly impaired". Higher scores indicate worsening.
Time Frame: Baseline, Day 14, Day 28, Day 42, and Day 56
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Escitalopram Oxalate
Number analyzed (Participants) | 234
Units on a scale
  Baseline (n=234) | 17.4 (5.87)
  Change at Day 14 (n=216) | -4.6 (5.80)
  Change at Day 28 (n=225) | -7.0 (6.09)
  Change at Day 42 (n=225) | -8.3 (6.73)
  Change at Day 56 (n=225) | -10.1 (6.80)

3. Secondary Outcome: Remission Rate Based on Montgomery-Asberg Depression Rating Scale (MADRS) up to Day 56
Description: Remission rate is defined as percentage of participants with MADRS total scores less than or equal to 10 at the endpoint (at week 8). The MADRS is a 10-item scale designed to measure depression severity. Each item is scored on 7-point scale, from 0 = not present/normal to 6 = severe/continuous presence of the symptoms and the total score (addition of all 10-items) ranges from "0 to 60". The interpretations of the scores are: 0 to 6= normal/symptom absent; 7 to 19= mild depression; 20 to 34= moderate depression; more than 34= severe depression.
Time Frame: Day 7, Day 14, Day 28, Day 42 and Day 56
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Escitalopram Oxalate
Number analyzed (Participants) | 240
Percentage of participants
  Day 7 (n=235) | 3.4 [1.1 to 5.7]
  Day 14 (n=240) | 16.3 [11.6 to 20.9]
  Day 28 (n=240) | 27.5 [21.9 to 33.2]
  Day 42 (n=240) | 43.3 [37.1 to 49.6]
  Day 56 (n=240) | 61.7 [55.5 to 67.8]

4. Secondary Outcome: Treatment Improvement Rate at the End of Week 1 and Week 2
Description: Onset of effect is defined as the reduction rate greater than or equal to 20 percent change from baseline in Montgomery-Asberg Depression Rating Scale (MADRS) total scores. The MADRS is a 10-item scale designed to measure depression severity. Each item is scored on 7-point scale, from 0 = not present/normal to 6 = severe/continuous presence of the symptoms and the total score (addition of all 10-items) ranges from "0 to 60". The interpretations of the scores are: 0 to 6= normal/symptom absent; 7 to 19= mild depression; 20 to 34= moderate depression; more than 34= severe depression.
Time Frame: Week 1 and Week 2
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Escitalopram Oxalate
Number analyzed (Participants) | 240
Participants
  Week 1 (n=235) | 98
  Week 2 (n=240) | 174

5. Secondary Outcome: Change in Montgomery-Asberg Depression Rating Scale (MADRS) Scores From Baseline up to Day 56
Description: The MADRS is a 10-item scale designed to measure depression severity. Each item is scored on a 7-point scale and the scores range from "0 = item not present/normal" to "6 = severe/continuous presence of the symptoms". Total score is calculated by adding the scores for all the 10 items and it ranges from "0 to 60". The interpretations of the scores are: 0 to 6= normal/symptom absent; 7 to 19= mild depression; 20 to 34= moderate depression; more than 34= severe depression.
Time Frame: Baseline, Day 7, Day 14, Day 28, Day 42 and Day 56
Population: Full Analysis Set Population included who received at least 1 dose of the study drug, and completed at least 1 assessment visit during the treatment period.
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Escitalopram Oxalate
Number analyzed (Participants) | 241
Units on a scale
  Baseline | 29.1 [28.2 to 29.9]
  Change at Day 7 | -5.6 [-6.4 to -4.9]
  Change at Day 14 | -10.5 [-11.5 to -9.5]
  Change at Day 28 | -13.6 [-14.7 to -12.5]
  Change at Day 42 | -16.4 [-17.6 to -15.3]
  Change at Day 56 | -19.1 [-20.2 to -17.9]

6. Secondary Outcome: Change in Hamilton Anxiety Scale (HAM-A) Total Scores From Baseline up to Day 56
Description: HAM-A is a rating scale developed to quantify the severity of anxiety symptomatology. It consists of 14 items, each defined by a series of symptoms. Each item is rated on a 5-point scale, ranging from 0 (not present) to 4 (severe). Total score is calculated by adding the scores for each of the 14 items and the score ranges from "0 to 56". The interpretation of total scores are: 0 to 17 is considered to be mild, 18 to 25 mild to moderate, and 26 to 30 moderate to severe and above 30 indicate very severe anxiety. Higher scores indicate worsening.
Time Frame: Baseline, Day 7, Day 14, Day 28, Day 42 and Day 56
Population: as for outcome 5
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Escitalopram Oxalate
Number analyzed (Participants) | 241
Units on a scale
  Baseline | 25.6 [24.7 to 26.5]
  Change at Day 7 | -5.6 [-6.4 to -4.8]
  Change at Day 14 | -10.1 [-11.1 to -9.1]
  Change at Day 28 | -12.9 [-13.9 to -11.9]
  Change at Day 42 | -15.1 [-16.2 to -14.0]
  Change at Day 56 | -17.5 [-18.6 to -16.4]

7. Secondary Outcome: Change in Inventory of Depressive Symptomatology, Self-Report (QIDS-SR) Total Scores From Baseline up to Day 56
Description: QIDS-SR contains 16 question regarding 9 Major depression disorder symptoms (sleep, weight, psychomotor changes, depressed mood, decreased interest, fatigue, guilt, concentration, and suicidal ideation). Each question is rated on a 4-point scale (range, 0 to 3). Total score is the sum of scores calculated by adding scores for each question and the interpretation is as follows: 0-5 (no depression likely); 6-10 (possibly mildly depressed); 11-15 (moderate depression); 16-20 (severe depression); 21-27 (very severe depression). Higher scores represent more severe depression symptoms.
Time Frame: Baseline, Day 7, Day 14, Day 28, Day 42 and Day 56
Population: as for outcome 5
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Escitalopram Oxalate
Number analyzed (Participants) | 241
Units on a scale
  Baseline | 14.9 [14.3 to 15.4]
  Change at Day 7 | -2.9 [-3.4 to -2.4]
  Change at Day 14 | -4.7 [-5.3 to -4.1]
  Change at Day 28 | -6.1 [-6.8 to -5.4]
  Change at Day 42 | -7.4 [-8.1 to -6.7]
  Change at Day 56 | -8.6 [-9.3 to -7.9]

8. Secondary Outcome: Depression Response Rate Based on Montgomery-Asberg Depression Rating Scale (MADRS) up to Day 56
Description: The MADRS is a 10 item scale designed to measure depression severity. Each item is scored on a 7 point scale and the scores range from "0 = item not present/normal" to "6 = severe/continuous presence of the symptoms". Total score is calculated by adding the scores for all the 10 items and ranges from "0 to 60". The interpretations of the scores are: 0 to 6= normal/symptom absent; 7 to 19= mild depression; 20 to 34= moderate depression; 35 to 60= severe depression data was obtained by Last observation carried forward (LOCF) method.
Time Frame: Day 7, Day 14, Day 28, Day 42 and Day 56
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Escitalopram Oxalate
Number analyzed (Participants) | 240
Percentage of participants
  Day 7 (n=235) | 7.2 [3.9 to 10.6]
  Day 14 (n=240) | 25.0 [19.5 to 30.5]
  Day 28 (n=240) | 46.7 [40.4 to 53.0]
  Day 42 (n=240) | 61.7 [55.5 to 67.8]
  Day 56 (n=240) | 74.2 [68.6 to 79.7]

9. Secondary Outcome: Remission Rate Based on Hamilton Anxiety Scale (HAM-A) up to Day 56
Description: HAM-A is a rating scale developed to quantify the severity of anxiety symptomatology. It consists of 14 items, each defined by a series of symptoms. Each item is rated on a 5 point scale, ranging from 0 (not present) to 4 (severe). Total score is calculated by adding the scores for each of the 14 items and the score ranges from "0 to 56". The interpretation of total scores are: 0 to 17 is considered to be mild, 18 to 25 mild to moderate, and 26 to 30 moderate to severe and 31 to 56 indicate very severe anxiety. Higher scores indicate worsening data was obtained by Last observation carried forward (LOCF) method.
Time Frame: Day 7, Day 14, Day 28, Day 42 and Day 56
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Escitalopram Oxalate
Number analyzed (Participants) | 240
Percentage of participants
  Day 7 (n=235) | 4.3 [1.7 to 6.8]
  Day 14 (n=240) | 15.8 [11.2 to 20.5]
  Day 28 (n=240) | 31.7 [25.8 to 37.6]
  Day 42 (n=240) | 43.8 [37.5 to 50.0]
  Day 56 (n=240) | 61.3 [55.1 to 67.4]

10. Secondary Outcome: Remission Rate Based on Inventory of Depressive Symptomatology, Self-Report (QIDS-SR) up to Day 56
Description: QIDS-SR contains 16 question regarding 9 Major depression disorder symptoms (sleep, weight, psychomotor changes, depressed mood, decreased interest, fatigue, guilt, concentration, and suicidal ideation). Each question is rated on a 4-point scale (range, 0 to 3). Total score is the sum of scores calculated by adding scores for each question and the interpretation is as follows: 0-5 (no depression likely); 6-10 (possibly mildly depressed); 11-15 (moderate depression); 16-20 (severe depression); 21-27 (very severe depression). Higher scores represent more severe depression symptoms data was obtained by Last observation carried forward (LOCF) method.
Time Frame: Day 7, Day 14, Day 28, Day 42 and Day 56
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Escitalopram Oxalate
Number analyzed (Participants) | 237
Percentage of participants
  Day 7 (n=228) | 7.5 [4.1 to 10.9]
  Day 14 (n=237) | 15.2 [10.6 to 19.8]
  Day 28 (n=237) | 27.0 [21.4 to 32.7]
  Day 42 (n=237) | 42.6 [36.3 to 48.9]
  Day 56 (n=237) | 51.5 [45.1 to 57.8]

ADVERSE EVENTS:
Time Frame: Baseline up to Day 56
Description: All participants who received at least 1 dose of the study drug were included in the Safety Analysis Set (SS). There were 257 participants included in the SS.
Arm/Group | Escitalopram Oxalate
Serious Adverse Events (participants affected / at risk) | 4/257
Other Adverse Events (participants affected / at risk) | 15/257
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Escitalopram Oxalate (N=257)
Suicide attempt (Psychiatric disorders) | 2
Hospitalisation (Surgical and medical procedures) | 1
Completed suicide (Psychiatric disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Escitalopram Oxalate (N=257)
Nausea (Gastrointestinal disorders) | 15 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.